CLINICAL TRIAL: NCT02993861
Title: Pharmacokinetics of Anti-epileptic Drugs in Obese Children
Status: Completed | Type: Observational
Sponsor: Christoph P Hornik, MD MPH (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Christoph P Hornik, MD MPH, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00070924
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Epilepsy; Obese
Keywords: Epilepsy; Obese
MeSH Terms: conditions — Epilepsy; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Levetiracetam: Children with epilepsy who are treated with levetiracetam per local standard of care
  Interventions: Other: Anti-epileptics
- Valproic Acid: Children with epilepsy who are treated with valproic acid per local standard of care
  Interventions: Other: Anti-epileptics
- Topiramate: Children with epilepsy who are treated with topiramate per local standard of care
  Interventions: Other: Anti-epileptics
- Oxcarbazepine: Children with epilepsy who are treated with oxcarbazepine per local standard of care
  Interventions: Other: Anti-epileptics

INTERVENTIONS:
Other: Anti-epileptics

SUMMARY:
The study is a prospective, multi-center, open-label clinical trial. Study's purpose is to characterize the pharmacokinetics and safety of four oral anti-epileptics drugs (levetiracetam, valproic acid [divalproex sodium ER or immediate release formulation if inadequate enrollment}, topiramate, and oxcarbazepine) in a non-randomized sample of obese children and adolescents. The study's duration will be up to eleven days (up to seven days of screening and four days of pharmacokinetic sampling). Eligible participants ages 2 to 18 years will be identified through outpatient clinic schedules and inpatient admissions at each clinic site. Participants receiving at least one of the study drugs per local standard of care will have pharmacokinetic concentrations in plasma drawn according to the specific dosing schedule for each drug. Other study measures include demographics, BMI, waist/hip ratio, medical history, concomitant medication history, documentation of study drug oral intake, adverse effects, and physical examination. The sample size will include 24 participants for each anti-epileptic drug (total 96).

ELIGIBILITY:
Inclusion Criteria:

* 2 years to < 18 years at the time of enrollment
* BMI ≥ 95th percentile for age and sex, based on CDC recommendations
* Informed consent/HIPAA from the parent/legal guardian and assent (as applicable)
* Receiving ≥ 1 of the study drugs per local standard of care

Exclusion Criteria:

* Known pregnancy as determined via interview or test results, if available

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with epilepsy who are inpatients in local hospital or managed in outpatient settings - community sample.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Steady-state pharmacokinetics area under the curve | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics maximum concentration | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics time to reach maximum concentration | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics oral apparent volume of distribution | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics half life | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics oral apparent clearance | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)
Steady-state pharmacokinetics absorption rate constant | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)

SECONDARY OUTCOMES:
Serious adverse events | Up to 14 days (up to 7 days of screening and 7 days of pharmacokinetic sampling)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, MPH, Principal Investigator — Duke Medical Center/Duke Clinical Research Institute
Locations (10):
- United States (10):
  - The Children's Hospital Colorado, Aurora, Colorado
  - Nemours Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Louisville Norton Childrens Hospital, Louisville, Kentucky
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Coastal Children's Services, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas